CLINICAL TRIAL: NCT01655212
Title: Congenital Cytomegalovirus: Efficacy of Antiviral Treatment in a Randomized Controlled Trial
Acronym: CONCERT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: 1 Indication for further investigations (brain ultrasound). 2 Change of study design to efficacy study with historical control group.
Sponsor: Dr. Ann C.T.M. Vossen (Other)
Collaborators: Stichting Nuts Ohra (Other); Leiden University Medical Center (Other)
Responsible Party: Sponsor-Investigator, Dr. Ann C.T.M. Vossen, MD, PhD, Dept of Medical Microbiology, Leiden University
Organization: Leiden University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMV-MM-1; 2011-005378-44 (EudraCT Number)
Record Dates: First submitted 2012-07-13; First posted 2012-08-01 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Congenital Cytomegalovirus Infection; Sensorineural Hearing Loss
Keywords: Cytomegalovirus; Congenital infection; Sensorineural hearing loss; Randomized controlled trial; Valganciclovir
MeSH Terms: conditions — Cytomegalovirus Infections; Hearing Loss, Sensorineural | interventions — Valganciclovir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Valganciclovir (Experimental): Valganciclovir 32 mg/kg per day in two doses (16 mg/kg per dose) during 6 weeks in an oral solution.
  Interventions: Drug: Valganciclovir
- Control (No Intervention): Infants in the control group receive no antiviral therapy. Counseling and treatment assigned by an audiological center remains unchanged.

INTERVENTIONS:
Drug: Valganciclovir — Infants will be treated with valganciclovir for 6 weeks, 32 mg/kg daily dose in two doses, oral solution.
  Other Names: Valcyte; Valganciclovirhydrochloride
  Arms: Valganciclovir

SUMMARY:
The objective of the trial is to investigate whether early treatment with oral valganciclovir of infants with both congenital cytomegalovirus infection and sensorineural hearing loss can prevent progression of hearing loss.

DETAILED DESCRIPTION:
In the Netherlands all neonates are routinely screened for hearing during the first weeks after birth with the Otoacoustic Emissions (OAE) procedure. After the second refer an Automated Auditory Brainstem Response (AABR) is performed. The parents of all newborns, born at ≥ 37 weeks gestational age, that fail this AABR in the Netherlands (about 550 yearly) will be asked for consent for CMV-testing on the dried blood spots. Newborns diagnosed with congenital CMV and with confirmed SNHL (≥ 20 dB) are eligible for inclusion. After informed consent infants will be randomized before the age of 13 weeks to a treatment group (6 weeks valganciclovir 32 mg/kg daily dose; oral solution) or control group (no antiviral treatment). Infants will be monitored for leucopenia and liver- and kidney function. Inclusion will continue for at least 1.5 years, or until 25 infants in each treatment arm have been randomized.

At 1 year follow-up hearing and child development are assessed. Hearing will be assessed with Brainstem Evoked Response Audiometry at an audiological center. Child development will be assessed during a home visit with the Bayley Scales of Infant Development III and parents will fill in the Dutch Child Development Inventory (NCDI) which will give more detailed information on communicative development of their child. Viral loads in blood and urine will be monitored during antiviral treatment as well as twice in the control group.

This study will provide information on the percentage of infants with a congenital CMV infection who fail the neonatal hearing screening . The RCT will show whether early treatment of congenital CMV infected children with hearing impairment prevents deterioration of hearing loss and to what extent. The outcome may lead to implementation of congenital CMV testing in the neonatal hearing screening program or possibly into the newborn blood screening.

ELIGIBILITY:
Inclusion Criteria:

* Infants with congenital CMV infection and hearing loss (≥ 20 dB, in one or both ears).
* Age at time of inclusion is < 13 weeks after birth.
* ≥ 37 weeks gestational age.
* Birth weight ≥ 2500 gram.
* Parental signed informed consent.

Exclusion Criteria:

* Indications for symptomatic congenital CMV infection based on diagnostics carried out prior to the inclusion of the child in the trial.
* In case during the house visit the presence of a symptomatic CMV infection is doubted, inclusion will be discussed. Depending on the medical history taking, physical examination and laboratory tests inclusion will be decided upon.
* Treatment with other antiviral agents or immunoglobulins.
* Leucopenia < 0,5 x 10*9/L (blood sample tested at t=0).

Ages: 3 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2012-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Hearing assessment | 1 year follow-up
  At 1 year follow-up hearing will be assessed with Brainstem Evoked Response Audiometry at an audiological center.

SECONDARY OUTCOMES:
Child development | 1 year follow-up
  At 1 year follow-up child development will be assessed during a home visit with the Bayley Scales of Infant Development III. Additionally, parents will fill in the Dutch Child Development Inventory.
Viral load | Baseline, weekly during 7 weeks, and at 1 year
  Viral blood load will be monitored in the treatment group(at baseline, weekly during antiviral treatment, and one week after treatment) as well as in the control group (baseline and 7 weeks after inclusion).
  Viral urine load will be monitored in the treatment group and in the control group (at baseline, weekly during 7 weeks after inclusion, and at the age of 1 year).

CONTACTS AND LOCATIONS:
Overall Officials: Ann CT Vossen, Dr., Study Director — Leiden University Medical Center; Anne Marie Oudesluys-Murphy, Prof. Dr., Principal Investigator — Leiden University Medical Center
Locations (1):
- Department Medical Microbiology, Leiden University Medical Center, Leiden, South Holland, Netherlands

REFERENCES:
- [Background] Kimberlin DW, Lin CY, Sanchez PJ, Demmler GJ, Dankner W, Shelton M, Jacobs RF, Vaudry W, Pass RF, Kiell JM, Soong SJ, Whitley RJ; National Institute of Allergy and Infectious Diseases Collaborative Antiviral Study Group. Effect of ganciclovir therapy on hearing in symptomatic congenital cytomegalovirus disease involving the central nervous system: a randomized, controlled trial. J Pediatr. 2003 Jul;143(1):16-25. doi: 10.1016/s0022-3476(03)00192-6. PMID 12915819
- [Background] Amir J, Wolf DG, Levy I. Treatment of symptomatic congenital cytomegalovirus infection with intravenous ganciclovir followed by long-term oral valganciclovir. Eur J Pediatr. 2010 Sep;169(9):1061-7. doi: 10.1007/s00431-010-1176-9. Epub 2010 Mar 16. PMID 20232081
- [Background] Lackner A, Acham A, Alborno T, Moser M, Engele H, Raggam RB, Halwachs-Baumann G, Kapitan M, Walch C. Effect on hearing of ganciclovir therapy for asymptomatic congenital cytomegalovirus infection: four to 10 year follow up. J Laryngol Otol. 2009 Apr;123(4):391-6. doi: 10.1017/S0022215108003162. Epub 2008 Jun 30. PMID 18588736
- [Background] Oliver SE, Cloud GA, Sanchez PJ, Demmler GJ, Dankner W, Shelton M, Jacobs RF, Vaudry W, Pass RF, Soong SJ, Whitley RJ, Kimberlin DW; National Institute of Allergy, Infectious Diseases Collaborative Antiviral Study Group. Neurodevelopmental outcomes following ganciclovir therapy in symptomatic congenital cytomegalovirus infections involving the central nervous system. J Clin Virol. 2009 Dec;46 Suppl 4(Suppl 4):S22-6. doi: 10.1016/j.jcv.2009.08.012. Epub 2009 Sep 18. PMID 19766534
- [Background] Michaels MG, Greenberg DP, Sabo DL, Wald ER. Treatment of children with congenital cytomegalovirus infection with ganciclovir. Pediatr Infect Dis J. 2003 Jun;22(6):504-9. doi: 10.1097/01.inf.0000069767.43169.2d. PMID 12799506
- [Background] Nigro G, Scholz H, Bartmann U. Ganciclovir therapy for symptomatic congenital cytomegalovirus infection in infants: a two-regimen experience. J Pediatr. 1994 Feb;124(2):318-22. doi: 10.1016/s0022-3476(94)70327-2. PMID 8301446
- [Background] Whitley RJ, Cloud G, Gruber W, Storch GA, Demmler GJ, Jacobs RF, Dankner W, Spector SA, Starr S, Pass RF, Stagno S, Britt WJ, Alford C Jr, Soong S, Zhou XJ, Sherrill L, FitzGerald JM, Sommadossi JP. Ganciclovir treatment of symptomatic congenital cytomegalovirus infection: results of a phase II study. National Institute of Allergy and Infectious Diseases Collaborative Antiviral Study Group. J Infect Dis. 1997 May;175(5):1080-6. doi: 10.1086/516445. PMID 9129069
- [Background] Smets K, De Coen K, Dhooge I, Standaert L, Laroche S, Mahieu L, Logghe N, Cossey V, Boudewyns A. Selecting neonates with congenital cytomegalovirus infection for ganciclovir therapy. Eur J Pediatr. 2006 Dec;165(12):885-90. doi: 10.1007/s00431-006-0192-2. Epub 2006 Jun 20. PMID 16786362
- [Background] Foulon I, Naessens A, Foulon W, Casteels A, Gordts F. A 10-year prospective study of sensorineural hearing loss in children with congenital cytomegalovirus infection. J Pediatr. 2008 Jul;153(1):84-8. doi: 10.1016/j.jpeds.2007.12.049. Epub 2008 Mar 6. PMID 18571542
- [Background] de Vries JJ, Korver AM, Verkerk PH, Rusman L, Claas EC, Loeber JG, Kroes AC, Vossen AC. Congenital cytomegalovirus infection in the Netherlands: birth prevalence and risk factors. J Med Virol. 2011 Oct;83(10):1777-82. doi: 10.1002/jmv.22181. PMID 21837795
- [Background] Korver AM, de Vries JJ, Konings S, de Jong JW, Dekker FW, Vossen AC, Frijns JH, Oudesluys-Murphy AM; DECIBEL collaborative study group. DECIBEL study: Congenital cytomegalovirus infection in young children with permanent bilateral hearing impairment in the Netherlands. J Clin Virol. 2009 Dec;46 Suppl 4:S27-31. doi: 10.1016/j.jcv.2009.09.007. PMID 19836301
- [Background] Fowler KB, McCollister FP, Dahle AJ, Boppana S, Britt WJ, Pass RF. Progressive and fluctuating sensorineural hearing loss in children with asymptomatic congenital cytomegalovirus infection. J Pediatr. 1997 Apr;130(4):624-30. doi: 10.1016/s0022-3476(97)70248-8. PMID 9108862
- [Background] Lanari M, Lazzarotto T, Venturi V, Papa I, Gabrielli L, Guerra B, Landini MP, Faldella G. Neonatal cytomegalovirus blood load and risk of sequelae in symptomatic and asymptomatic congenitally infected newborns. Pediatrics. 2006 Jan;117(1):e76-83. doi: 10.1542/peds.2005-0629. Epub 2005 Dec 1. PMID 16326692
- [Background] Lombardi G, Garofoli F, Stronati M. Congenital cytomegalovirus infection: treatment, sequelae and follow-up. J Matern Fetal Neonatal Med. 2010 Oct;23 Suppl 3:45-8. doi: 10.3109/14767058.2010.506753. PMID 20807160
- [Background] Misono S, Sie KC, Weiss NS, Huang ML, Boeckh M, Norton SJ, Yueh B. Congenital cytomegalovirus infection in pediatric hearing loss. Arch Otolaryngol Head Neck Surg. 2011 Jan;137(1):47-53. doi: 10.1001/archoto.2010.235. PMID 21242546
- [Background] Kimberlin DW, Acosta EP, Sanchez PJ, Sood S, Agrawal V, Homans J, Jacobs RF, Lang D, Romero JR, Griffin J, Cloud GA, Lakeman FD, Whitley RJ; National Institute of Allergy and Infectious Diseases Collaborative Antiviral Study Group. Pharmacokinetic and pharmacodynamic assessment of oral valganciclovir in the treatment of symptomatic congenital cytomegalovirus disease. J Infect Dis. 2008 Mar 15;197(6):836-45. doi: 10.1086/528376. PMID 18279073